CLINICAL TRIAL: NCT04029181
Title: ImmunoPET Imaging With ZED88082A in Patients Before and During Treatment With 1) MPDL3280A or 2) PD-1 Antibody Plus or Minus Ipilimumab
Brief Title: ImmunoPET With an Anti-CD8 Imaging Agent
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201700848
Record Dates: First submitted 2019-06-17; First posted 2019-07-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Cancer; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose finding cohort (Experimental): In part A of this imaging trial, a dose finding study will be performed to establish safety, to assess the appropriate protein dose for PET-scanning and to assess the appropriate PET scanning interval.
  Interventions: Other: Anti-CD8 PET imaging agent
- Feasibility cohort (Experimental): The purpose of part B of the study is to analyze the PK of the anti-CD8 imaging agent in patients before and during treatment with checkpoint inhibitors.
  Interventions: Other: Anti-CD8 PET imaging agent

INTERVENTIONS:
Other: Anti-CD8 PET imaging agent — An imaging agent radiolabelled with 89Zr developed for in human PET imaging of CD8

SUMMARY:
This is a single-center, single-arm, investigator sponsored trial designed to evaluate the PK of the anti-CD8 imaging agent in patients prior to and during treatment with checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed locally advanced or metastatic cancer for the following tumor types

   * Cancer types other than melanoma; subjects meeting the eligibility criteria as formulated in the MPDL3280A treatment study protocol (MPDL3280A-treatment-IST-UMCG) are eligible for part A or part B1.
   * Melanoma; subjects eligible to receive standard of care anti-PD1 therapy plus or minus ipilimumab, are eligible for part B2.
2. Tumor lesion(s) of which a histological biopsy can safely be obtained according to standard clinical care procedures.
3. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions.
4. Signed informed consent.
5. Age ≥18 at the time of signing informed consent.
6. Life expectancy ≥12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Ability to comply with the protocol.
9. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly).

Exclusion Criteria:

1. Potential subjects with cancer other than melanoma will be excluded from participation in this study if they meet exclusion criteria formulated in the MPDL3280A treatment study protocol (MPDL3280A-treatment-IST-UMCG).
2. Signs or symptoms of infection within 2 weeks prior to anti-CD8 imaging agent injection.
3. Prior immune checkpoint inhibitor treatment, including but not limited to anti-PD1 and anti-PD-L1 therapeutic antibodies.
4. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
5. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the anti-CD8 imaging agent, or that may affect the interpretation of the results or render the patient at high risk from complications.
6. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events related to tracer administration as assessed by CTCAE v4.0 | 2 years
  Safety assessment through summaries of adverse events, changes in laboratory test results (if evaluation is indicated), changes in vital signs, and exposure to ZED88082A/CED88004S. Adverse event data will be recorded and summarized according to NCI CTCAE v4.0.
Appropriate dosing of anti-CD8 imaging agent and PET imaging time points | 2 years
  Appropriate dosing and imaging time points of the anti-CD8 imaging agent will be determined based on measurements of standardized uptake value (SUV) of defined volumes of interest (VOIs) on the immunoPET scan images
Pharmacokinetics (PK) of anti-CD8 imaging agent | 2 years
  Description of PK of the anti-CD8 imaging agent by measuring standardized uptake value (SUV) on PET scans performed 0, 2, 4 and/or 7 days after tracer injection before and during MPDL3280A or PD-1 antibody immune checkpoint inhibitor plus or minus ipilimumab treatment.
Immunogenic potential of the anti-CD8 imaging agent by measuring incidence of anti-drug antibodies | 2 years
  Assessment of the immunogenic potential of the anti-CD8 imaging agent by measuring incidence of anti-drug antibodies during the study relative to the prevalence of ADAs at baseline and assessing their relationship to other outcomes measured.

SECONDARY OUTCOMES:
Heterogeneity of tumor uptake of the anti-CD8 imaging agent | 2 years
  Heterogeneity of imaging tracer uptake will be evaluated by measuring standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the immunoPETscan images
Correlation of normal organ uptake of the anti-CD8 imaging agent to (serious) adverse events (possibly) related to immune checkpoint inhibitor treatment | 2 years
  Normal organ uptake of the anti-CD8 imaging agent as measured by SUVs on PET scan images will be analyzed on correlation to (serious) adverse events (possibly) related to ICI treatment, defined as all (S)AEs which are assessed as "possibly", "probably" or "definitely" related to ICI treatment.
Correlation of tumor uptake of the anti-CD8 imaging agent and immune cell CD8 expression | 2 years
  Results of immunohistochemical scoring of tumor and immune cell CD8 and other markers of lymphocytic infiltration in fresh biopsies will be described as a semi-quantitative score using the percentage of positive cells (continuous variable), intensity and pattern of staining (discrete variable). These IHC results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the immunoPETscan images. Results of autoradiography will be described by measuring standardized uptake value (SUV) on the biopsy slides.
Correlation of anti-CD8 imaging agent normal tissue kinetics with blood kinetics | 2 years
  PK parameters will be derived from anti-CD8 imaging agent serum concentrations and will be summarized using descriptive statistics including but not limited to the number of patients, mean, standard deviation, median, minimum and maximum.
Dosimetry | 2 years
  Assessment of dosimetry will be performed by calculations of radioactivity in Bq or mSv of anti-CD8 imaging agent concentration in tumor target tissue, blood and other organs of interest with regards to injected dose (ID), derived from measurements of standardized uptake value (SUV) on immunoPET images and direct analysis of blood 89Zr-activity.

CONTACTS AND LOCATIONS:
Overall Officials: E. G.E. de Vries, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Kist de Ruijter L, van de Donk PP, Hooiveld-Noeken JS, Giesen D, Elias SG, Lub-de Hooge MN, Oosting SF, Jalving M, Timens W, Brouwers AH, Kwee TC, Gietema JA, Fehrmann RSN, Fine BM, Sanabria Bohorquez SM, Yadav M, Koeppen H, Jing J, Guelman S, Lin MT, Mamounas MJ, Eastham JR, Kimes PK, Williams SP, Ungewickell A, de Groot DJA, de Vries EGE. Whole-body CD8+ T cell visualization before and during cancer immunotherapy: a phase 1/2 trial. Nat Med. 2022 Dec;28(12):2601-2610. doi: 10.1038/s41591-022-02084-8. Epub 2022 Dec 5. PMID 36471036
- [Derived] Ogasawara A, Kiefer JR, Gill H, Chiang E, Sriraman S, Ferl GZ, Ziai J, Bohorquez SS, Guelman S, Wang X, Yang J, Phan MM, Nguyen V, Chung S, Yu C, Tinianow J, Waaijer SJH, De Crespigny A, Marik J, Boswell CA, Zabka T, Staflin K, Williams SP. Preclinical development of ZED8, an 89Zr immuno-PET reagent for monitoring tumor CD8 status in patients undergoing cancer immunotherapy. Eur J Nucl Med Mol Imaging. 2023 Jan;50(2):287-301. doi: 10.1007/s00259-022-05968-6. Epub 2022 Oct 22. PMID 36271158